CLINICAL TRIAL: NCT04309903
Title: The Effectiveness of Manual Theraphy on Lower Extremity Joint Arthropathy in Patients With Hemophilia
Brief Title: The Effects of Manual Therapy in Hemophilic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Necati Muhammed TAT, Lecturer, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Necmettin Erb. Physiotherapy-2
Record Dates: First submitted 2020-03-13; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Hemophilia; Arthropathy Hemophilic
Keywords: Hemophilia; Arthropathy; Physiotherapy; Manual therapy; Joint health
MeSH Terms: conditions — Hemophilia A; Joint Diseases | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Therapy (Experimental): The experienced physiotherapist has applied manual therapy (MT) to the arthropathic joints. MT was started with myofascial release techniques (MRT), then continued with mobilization techniques using Kalternborn. Superficial MRT consisted of 3 strokes, via manual movement on the tissue, encourage release of the superficial fascia. In the Kalternborn mobilization technique, Grade I-II mobilization was applied with traction without using a strap. The same exercises given to the home exercise group were given to the patients in this group as well.
  Interventions: Other: Manual therapy
- Home Exercise (Active Comparator): The home exercises (HE) consisted of active ROM exercises, passive stretching exercises, progressive resistive exercises, weigh-bearing and stance exercises were performed by the patient for 30 minutes at home.
  Interventions: Other: Manual therapy

INTERVENTIONS:
Other: Manual therapy — Both groups received for 3 sessions per week, a total of 5 weeks. Home exercises were performed by the patient for 30 minutes at home.In home exercises active ROM for warm-up (5 min), passive stretchening (5 min), strengthening exercises (10 min), proprioceptive and balance exercises (10 min). In manual therapy group, myofascial release techniques (MRT) and Kalternborn mobilization techniques lasted about one hour. In MRT, each manuever was applied for 2 mins and 3 times. The superficial strokes were performed, assisted by slight movements of joints. MRT to posterior capsule of the knee, ligaments, iliotibial tractus, plantar fascia, metatarsal, tarsals, and toes. Kalterborb mobilization tecnqiues; posterior gliding for restricted knee flexion, anterior gliding for restricted knee extension,talocrural posteior gliding for dorsal flexion, talocrural anterior gliding for plantar flexion.3 * 10 repetitions, 20 sec of per reps and 10 sec of interval.
  Other Names: Home exercise

SUMMARY:
Uncertainty about how to treat existing hemophilic arthropathy (HA) is the most important issue that will increase functionality and joint health. Recent studies have shown that MT can be used safely for improving joint health, pain and ROM with no bleedings in PwH with elbow and ankle HA. Unlike MT studies in hemophilia, we investigated the effects of MT on important parameters such as muscle strength (MS), functional level, joint health, functional independence score in hemophilia (FISH) and kinesiophobia. These parameters are closely related to functional level and quality of life of PwH. Therefore, evaluation of these parameters and determining the effects of the MT on these parameters are very important for both PwH and also clinicians.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effects of manual therapy in addition to home exercise program on hemophilia functional independence level, joint health, kinesiophobia, functional level, range of motion, muscle strength and pain level in hemophilic individuals with lower extremity joint arthropathy. Hemophilic arthropathy was developed in at least one of the lower extremity joints and aged between 18-30 years 17 severe type hemophilic men were participated in the study. The participants were divided into two groups as Home Exercise Group (HEG) and Manual Therapy Group (MTG) by randomization method. While the HEG was performed the exercise program at home, in addition to the same HEG manual therapy were applied to the MTG by the same physiotherapist 3 days a week for 1 hour. Both groups were followed for a total of 5 weeks and pre-treatment evaluations were repeated post-treatment. The joint health of the hemophilics in both groups were evaluated with Hemophilia Joint Health Score (HJHS), their kinesiophobia level were evaluated with Tampa Kinesophobia Scale, their functionality with the Functional Independence Score in Hemophilia (FISH). In addition, Functional Reach, Timed Up and Go and 5 Times Sit-to- Stand tests were used for functional level. The range of motion was evaluated with a goniometer, muscle strength was measured with a digital dynamometer and pain level was assessed with a Visual Analogue Scale (VAS). Number of hemarthrosis decreased in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemophilia who have arthropathy developed in any of the lower extremity joints due to severe hemophilia and to be receiving regular prophylaxis (3*1500 IU/ per week), but not having regular physical activity and sports.

Exclusion Criteria:

* Patients with hemophilia who had any disease related to connective tissue, any surgery that affects lower limb function (joint debridement, fracture, prosthesis), any neurological disease or cognitive impairment that may affect functional level, any sensorial loss of peripheral nerve injury and did not attend their sessions and evaluations regularly.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
Hemophilia Joint Health Score | 5 week
  We used the index point of joints. Score ranged from 0 to 20. Low score indicates the good joint health
Functional Independence Score in Hemophilia | 5 week
  We used the functional independence of patients. Score ranged from 0 to 32. High score indicates the functional independence.
Tampa Kinesiophobia Scale | 5 week
  Score higher than 37 were associated with a high degree of kinesiophobia.

SECONDARY OUTCOMES:
Range of motion | 5 week
  Joint range was measured with a universal goniometer.
Muscle Strength | 5 week
  It was measured with hand-held dynamometer.
Numerical Pain Scale | 5 week
  It was used for assessment of activity and resting pain.
Frequency bleeding | 5 week
  It was evaluated from the diaries kept by the patients
Functional Reach | 5 week
  It was used to assess dynamic balance.
Timed Up and Go | 5 week
  It was used to evaluate functional mobility, dynamic balance, fall risk and postural stability.
5 Times Sit to Stand | 5 week
  It was evaluated the functional strength of lower extremity, transitive movements, balance and fall risk.

CONTACTS AND LOCATIONS:
Overall Officials: Filiz CAN, Professor, Study Chair — Hacettepe University, Faculty of Physiotherapy and Rehabilitation; Ilgen SASMAZ, Professor, Study Director — Cukurova University; Ali Bulent ANTMEN, Professor, Study Director — Acıbadem Adana Hospital
Locations (1):
- Cukurova University, Adana, Sarıcam, Turkey (Türkiye)